CLINICAL TRIAL: NCT07007624
Title: Basketball Intervention Program In Children
Acronym: BIPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIPIC
Record Dates: First submitted 2025-05-05; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Basketball
Keywords: Basketball; Inflammation; Sports; Health; Childhood; Diet
MeSH Terms: conditions — Inflammation | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basketball training (Sport and diet) (Experimental)
  Interventions: Other: Basketball training (Sport and diet)

INTERVENTIONS:
Other: Basketball training (Sport and diet) — The intervention program will last for 3 years, and each year will be divided into two periods: a preseason, beginning in early September and lasting for the first 6 weeks, followed immediately by a 32-week season (until the end of the school year). The preseason will include 5 training sessions per week, each lasting 2 hours (Monday to Friday). The following season will include 3 training sessions per week, each lasting 2 hours (after school), and one match on the weekend. Each session will be divided into 2 periods separated by a 10-minute break: the first period will focus on individual skills with moderate to high-intensity exercises (60-85% of heart rate), and the second period will focus on gameplay (tactics and strategy). The trainers had a high level of professional training, ensuring the quality of the sessions. Dietary recommendations based on the Mediterranean diet will be given to the subjects.

SUMMARY:
The current project is a longitudinal, clinical study focused on evaluating the effects of a structured physical activity intervention in healthy prepubertal boys. The study will be conducted with the collaboration of the Pediatrics Department and the Nutrition and Metabolism Area of the Reina Sofía University Hospital in Córdoba; the Child Metabolism and Nutrigenomics. Metabolic Syndrome research groups at the Maimónides Institute for Biomedical Research (IMIBIC); and the Departments of Biochemistry at both the University of Córdoba and the University of Granada.

A total of 20 male participants, aged 9 to 12 years, will be selected. Inclusion criteria include being healthy, in Tanner stage I of pubertal development, and having anthropometric and cardiovascular parameters (weight, height, BMI, heart rate, systolic and diastolic blood pressure) within the 50th percentile ±1 standard deviation. Children outside this range, or with signs of pubertal development, will be excluded.

The intervention consists of a 3-year physical activity program structured into two annual phases: a 6-week preseason beginning each September, followed by a 32-week season coinciding with the academic year. During the preseason, participants will undergo five weekly 2-hour training sessions. The season will include three 2-hour after-school training sessions per week, and one weekend match. Training sessions will be divided into two parts: individual skill development at moderate to high intensity (60-85% HR) and gameplay focusing on tactics and strategy. All sessions will be supervised by highly qualified coaches.

Physical fitness will be assessed through the Eurofit test battery, including the Course Navette, Sit and Reach, 30-second Sit-ups, and Standing Long Jump tests. Physical activity levels will be monitored using accelerometers, and data on weekly activity frequency, intensity, sedentary behavior, and leisure time will be collected. A comprehensive physical examination will include assessment of pubertal development, anthropometry, heart rate, and blood pressure. Body composition will be measured using TANITA BC-418 bioimpedance equipment, and will include height, weight, lean and fat mass, and body water percentage. Additionally, biochemical markers of general health, inflammation (via LINCOplex assays and Luminex xMAP technology), and oxidative stress will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male children
* Weight, height, BMI, heart rate, systolic and diastolic blood pressure within the 50th percentile ±1 SD
* Tanner stage I of pubertal development

Exclusion Criteria:

* Boys younger than 9 or older than 12 years
* Anthropometric or physiological values above the 75th or below the 25th percentile

Ages: 9 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Body composition: Height | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Height in centimeters is measured with the SECA 213 precision measuring instrument on an annual basis.
Body composition: Weight | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Weight in grams is measured by the precision weighing scale model Tanita 780PMA on an annual basis.
Body composition: Body mass index | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Body mass index in kilograms per square meter is calculated on an annual basis.
Body composition: Waist circumference | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Waist circumference in centimeters is measured with a SECA 201 precision measuring tape on an annual basis.
Muscular strength | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  The upper and lower body strength was assayed by the flexed arm hang (FAH) and horizontal jump test, quantifying the time maintaining a flexion and the distance reached in the jumps, respectively
Cardiorespiratory endurance | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Cardiorespiratory endurance is assessed in minutes by using the Course Navette test. The number of completed series is recorded.
Anaerobic capacity | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Core strength was evaluated by the number of abdominals in 30 seconds
Anaerobic capacity | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Anaerobic capacity was assessed by the speed test (40 m)

SECONDARY OUTCOMES:
Assessment of dietary intake and habits | September, January, April, and June of the first year, September of the second year, and September of the third year.
  The habitual intake of the child is assessed by using the food and drink frequency questionnaire and KID-MED.
  The KIDMED index ranges from -4 to 12 points. Higher scores indicate greater adherence to the Mediterranean diet and therefore a better dietary quality. A total score is calculated based on 16 yes/no questions: positive connotations are scored +1, and negative connotations are scored -1.
Body composition: Fat mass | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Fat mass both in kilograms and in percentage is measured on an annual basis.
Body composition: Fat mass index | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  Fat mass index in kilograms per square meter is calculated on an annual basis.
Body composition: Fat-free mass | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Fat-free mass in kilograms is measured on an annual basis.
Body composition: Total body water | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Total body water both in kilograms and in percentage is measured on an annual basis.
Systolic blood pressure measurement | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  On an annual basis, the systolic blood pressure is measured in mmHg in triplicate in order to obtain an average value.
Diastolic blood pressure measurement | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  On an annual basis, the diastolic blood pressure is measured in mmHg in triplicate in order to obtain an average value.
Heart rate measurement | In the first year, measurements were taken at baseline (September), and at 6, 9, and 12 months. In the third year, the same measurement schedule was repeated.
  On an annual basis, the heart rate is measured in beats per minute in triplicate in order to obtain an average value.
Hematological analysis: Hemoglobine | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Hemoglobin levels are determined in grams per deciliter on an individual basis.
Hematological analysis: Hematocrite | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Hematocrite levels are determined in percentage on an individual basis.
Hematological analysis: Erythrocytes | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Erythrocytes count is measured in 10e06 units per microliter on an individual basis.
Hematological analysis: Mean corpuscular volume | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Mean corpuscular volume is measured in femtoliters on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Mean corpuscular hemoglobine is measured in picograms on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin concentration | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Mean corpuscular hemoglobine concentration is measured in grams per deciliter on an individual basis.
Hematological analysis: Red cell blood distribution width | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Red cell blood distribution width is determined in percentage on an individual basis.
Hematological analysis: White blood cells | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.ual basis.
  White blood cells count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Neutrophils | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Neutrophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Lymphocytes | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Lymphocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Monocytes | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Monocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Eosinophils | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Eosinophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Basophiles | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Basophiles count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Platelets | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Platelets count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Mean platelet volume | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Mean platelet volume is measured in femtoliters on an individual basis.
Biochemical analysis: Glucose | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Glucose is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Bilirubin | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Total bilirubin is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Creatinine | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Creatinine is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urate | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Urate is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urea | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Urea is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total protein | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Total protein is measured both in grams per deciliter and in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Aspartate aminotransferase | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Aspartate aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alanine aminotransferase | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Alanine aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Gamma-glutamyl transferase | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Gamma-glutamyl transferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alkaline phosphatase | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Alkaline phosphatase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total cholesterol | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Total cholesterol is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: High density lipoproteins | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  High density lipoproteins (HDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Non-HDL cholesterol | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Non-HDL cholesterol levels are calculated in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Low density lipoproteins | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Low density lipoproteins (LDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein A1 | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Apolipoprotein A1 is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein B | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Apolipoprotein B is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Calcium | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Calcium is measured both in milligrams per deciliter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Potassium | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Potassium is measured both in millimoles per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sodium | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Sodium is measured in millimoles per liter, in milliequivalents per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Phosphorus | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Phosphorus is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Iron | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Iron is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Magnesium | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Magnesium is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Zinc | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Zinc is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Insulin is measured both in micro international units per liter and in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin resistance | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) index is used to estimate insulin resistance.
Biochemical analysis: C-reactive protein | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  C-reactive protein is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Tumor necrosis factor alpha | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Tumor necrosis factor alpha is measured in picograms per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Adiponectin | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Adiponectin is measured in milligrams per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: IL-6 | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Il-6 is measured in picograms per milliliter on an individual basis. Analysis performed in plasma.
IL-8 | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  IL-8 is measured in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: NGF | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  NGF is measured in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: TNFa | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  TNFa is measured in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: MCP-1 | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  MCP-1 is measured in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total PAI-1 | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  Total PAI-1is measured in units per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: HGF | Measurements were taken at baseline in September and 9 months later in June during the first year. This same schedule was repeated in the third year.
  HGF is measured in nanograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Energy | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Energy is determined in kilocalories on an individual basis. Analysis performed in plasma.
Biochemical analysis: Carbohydrates | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Carbohydrates are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sugars | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Sugars are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Fiber | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Fibers are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polysaccharides | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Polysaccharides are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total fat | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Total fat is measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Saturated fatty acids | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Saturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Monounsaturated fatty acids | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Monounsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polyunsaturated fatty acids | September, January, April, and June of the first year, September of the second year, and September of the third year.
  Polyunsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- IMIBIC, Córdoba, Spain

REFERENCES:
- [Derived] Castro-Collado C, Jurado-Castro JM, Gil-Campos M, Cruz Rico M, Pastor-Villaescusa B, Quintana-Navarro GM, Llorente-Cantarero FJ. Changes in body composition and low-grade inflammation status in boys during a basketball afterschool program for three years. Sci Rep. 2025 Nov 6;15(1):38916. doi: 10.1038/s41598-025-22628-5. PMID 41198734
- [Derived] Castro-Collado C, Jurado-Castro JM, Gil-Campos M, Pastor-Villaescusa B, Quintana-Navarro GM, Llorente-Cantarero FJ. Effects of After-School Basketball Program on Physical Fitness and Cardiometabolic Health in Prepubertal Boys. Sports (Basel). 2025 Aug 28;13(9):291. doi: 10.3390/sports13090291. PMID 41003597